CLINICAL TRIAL: NCT01136902
Title: Measuring Retinal Vessel Caliber in Relation to Dark Adaptation and Blood Glucose Level
Status: Completed | Type: Observational
Sponsor: Glostrup University Hospital, Copenhagen (Other)
Responsible Party: Stig Holfort, MD, Glostrup University Hospital,Copenhagen
Other Study IDs: Kappelgaard, vessel
Record Dates: First submitted 2010-06-01; First posted 2010-06-04 (Estimated); Last update posted 2010-12-08 (Estimated); Status verified 2010-12

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes Mellitus; Retinal Vessels; Physiology
MeSH Terms: conditions — Diabetes Mellitus | interventions — Glucose Tolerance Test

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Venous blood sample. Na+, K+, Crea, HbA1c. Capillary glucose measurement. Samples will be analysed and destructed according to normal laboratory practice at the Glostrup Hospital.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Type 2 DM: This group includes subjects diagnosed with type 2 diabetes mellitus with none or minimal diabetic retinopathy.
  Interventions: Dietary Supplement: Oral Glucose Tolerance Test (OGTT)

INTERVENTIONS:
Dietary Supplement: Oral Glucose Tolerance Test (OGTT) — 75 g of glucose dissolved in 250 mL water.
  Other Names: OGTT

SUMMARY:
The overall objective is to investigate, whether retinal blood vessel diameter change during the energy consuming dark adaptation process and if responses vary between low and high blood glucose.

DETAILED DESCRIPTION:
All subjects are being studied using the same procedure. The study schedule takes place from 8 a.m. to 12 a.m. every time. Each subject shows up on one single day. Subjects are to show up fasting overnight with a break in insulin and/or oral antidiabetic treatment.

The study eye of each subject will be selected by randomisation. We seek to have an equal distribution of right and left eyes overall.

A first set of images will be taken after 5 minutes in "standardised daylight", in a room without light from outside, which eliminates any concerns about weather variations. After this the room is completely darkened. 2 set of images will be taken in the dark adapted state after 20 and 40 minutes. Subsequently the patient ingests the OGTT and will reach maximum blood glucose level after about 60-90 minutes. At this time, the subjects undergo the same "photo session" as above with high blood glucose levels.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetic individuals.
* minimal or no diabetic retinopathy defined by no more than five microaneurysms or dot hemorrhages per eye on three non-stereoscopic 50 degree color fundus photographs

Exclusion Criteria:

* Test individuals with significant cataract, prior surgery to the eye, diabetic retinopathy, other serious eye disease, hypertension, other serious systemic disease

Ages: 17 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects with diagnosed Type 2 diabetes mellitus with none or minimal diabetic retinopathy.
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2009-08; Primary Completion 2010-06 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Vessel caliber | 1 day

SECONDARY OUTCOMES:
Blood glucose level | 1 day
  Capillary samples.

CONTACTS AND LOCATIONS:
Overall Officials: Stig K Holfort, MD, Principal Investigator — Glostrup University Hospital, Copenhagen
Locations (1):
- Copenhagen University Hospital at Glostrup, Copenhagen, Copenhagen, Denmark